CLINICAL TRIAL: NCT02070640
Title: Near Infrared Fluorescence Cholangiography During Cholecystectomy
Brief Title: Near Infrared Fluorescence Cholangiography (NIRF-C) During Cholecystectomy
Acronym: NIRF-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Stryker Instruments (Industry); Society of American Gastrointestinal and Endoscopic Surgeons (Other)
Responsible Party: Principal Investigator, Narula, Vimal K, MD, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011H0239
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Cholecystitis
Keywords: cholecystectomy; cholecystitis
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NIRF-C (Experimental): Each subject enrolled in this study will undergo near-infrared cholangiography fluorescence (NIRF-C) and standard of care intraoperative cholangiography. 2.5 mg of indocyanine green is injected 30-60 minutes prior to surgery. Visualization of the biliary tree during surgery is achieved with a near-infrared light source and camera.
  Interventions: Drug: Injection of indocyanine green (ICG); Device: Near Infrared Cholangiography Fluorescence (NIRF-C)

INTERVENTIONS:
Drug: Injection of indocyanine green (ICG) — 2.5 mg of of ICG will be injected intravenously 60-30 minutes prior to surgery in order to visualize the biliary tree using a near-infrared light source and camera. An additional 2.5 mg of IV ICG may be given intraoperatively if fluorescence has faded prior to visualization.
Device: Near Infrared Cholangiography Fluorescence (NIRF-C) — These devices are used to identify anatomy, using infrared light that causes the ICG to fluoresce.
  Other Names: Stryker 1488 Camera System; Stryker L9000 Light Source; Stryker 1488 Coupler; Stryker 10mm Ideal Eyes Laparoscope (0 and 30 degree)

SUMMARY:
The purpose of this study is to evaluate an imaging system using Indocyanine Green (ICG) to assist in real-time identification of anatomy during cholecystectomy (gallbladder removal). We propose to define the effectiveness of NIRF-C in identifying the cystic duct junction during cholecystectomy.

DETAILED DESCRIPTION:
This study is designed to determine the clinical utility of intravenous indocyanine green (ICG) injection pre-operatively for cholecystectomy, followed by visualizuation of the biliary tree with a near-infrared light source and camera. Testing will be done during an abdominal surgery which requires gallbladder removal. Subjects will be recruited during consult for their surgical procedure. The study itself will take an estimated 5 minutes during the procedure. 2.5mg of ICG will be injected intravenously 60-30 minutes before surgery, and following perfusion of the biliary tree, images will be recorded and visibility of the appropriate anatomy will be assessed using a near-infrared light source and camera. If fluorescence has faded prior to adequate visualization, a repeat dose of 2.5mg IV ICG may be given. Following the completion of imaging, the standard procedure for cholecystectomy will be performed including intraoperative cholangiography (IOC), which is standard of care. Subject post-operative recovery will be monitored for the duration of their hospital stay. Adverse events will be monitored at the patient's routine follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Planned laparoscopic cholecystectomy

Exclusion Criteria:

* Inability to provide informed consent
* Pregnant
* Allergy to ICG, iodine, and/or shellfish
* Acute cholecystitis, cholangitis, and/or cirrhosis (main study)
* Lactating

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vimal K Narula, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-acute; Acute Cholecystitis: Each subject enrolled in this study will undergo near-infrared cholangiography fluorescence (NIRF-C) and standard of care intraoperative cholangiography.
  Injection of indocyanine green (ICG): 2.5 mg of of ICG will be injected intravenously 60-30 minutes prior to surgery. An additional 2.5 mg of IV ICG may be given intraoperatively if fluorescence has faded prior to visualization.
  Near Infrared Cholangiography Fluorescence (NIRF-C): These devices are used to identify anatomy, using infrared light that causes the ICG to fluoresce.
Period: Overall Study
Arm/Group | Non-acute | Acute Cholecystitis
Started | 93 | 6
Completed | 82 | 6
Not Completed | 11 | 0

BASELINE CHARACTERISTICS:
Population: Cholecystitis or acute cholecystitis
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Acute | Acute Cholecystitis | Total
Number analyzed (Participants) | 82 | 6 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 6 | 84
  >=65 years | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 3 | 67
  Male | 18 | 3 | 21
Region of Enrollment [Number; unit: participants]
  United States | 82 | 6 | 88

OUTCOME MEASURES:

1. Primary Outcome: Complications Related to ICG
Description: A patient's negative reaction to indocyanine green (ICG) will be monitored from the time of injection through the 2 week post-operative follow-up visit.
Time Frame: From time of injection to 1st post-op follow-up
Measure: Number; unit: % of Participants with Complications
Arm/Group | Non-Acute | Acute Cholecystitis
Number analyzed (Participants) | 82 | 6
% of Participants with Complications | 0 | 0

2. Secondary Outcome: Incidence of Anatomic Identification With NIRF-C
Description: Incidence of anatomic identification with NIRF-C and intraoperative cholangiography.
Time Frame: Intraoperative
Measure: Number; unit: percentage of biliary anatomy observatio
Arm/Group | Non-Acute | Acute Cholecystitis
Number analyzed (Participants) | 82 | 6
percentage of biliary anatomy observatio | 95.1 | 33

3. Secondary Outcome: Time to Complete NIRF-C and IOC
Description: The time required to complete NIRF-C and intraoperative cholangiography will be analyzed.
Time Frame: Intraoperative
Measure: Mean (Full Range); unit: minutes
Arm/Group | Non-acute | Acute Cholecystitis
Number analyzed (Participants) | 82 | 6
minutes | 1.9 [.2 to 3.6] | 1.08 [.25 to 1.28]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Non-acute | Acute Cholecystitis
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/6
Other Adverse Events (participants affected / at risk) | 1/93 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-acute (N=93) | Acute Cholecystitis (N=6)
IV infiltration of ICG (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes